CLINICAL TRIAL: NCT06327997
Title: Exploratory Study on the Treatment of Advanced Solid Tumor With Non-viral Vector Multi-targeted Autosecretory Multifunctional Antibody CAR-T Cell Injection
Brief Title: An Exploratory Study by Fast CAR T Cells
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZE2203-A-01
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fast CAR T cells (Experimental): Pretreatment was given 5 days before CAR T infusion for 3 consecutive days, and CAR T cell infusion was performed on the 0th day
  Interventions: Biological: Fast CAR T cells

INTERVENTIONS:
Biological: Fast CAR T cells — This study designed three dose groups, each with a dosage of 5.0 × 10^5/kg、1.0×10^6/kg、5.0×10^6/kg

SUMMARY:
The main goal of this trial is to evaluate the safety and tolerability of CAR T cell therapy for advanced solid tumors with positive mesothelin and MUC1.Patients were screened, peripheral blood mononuclear cells (PBMC) were isolated from eligible patients, and cells were prepared. Pretreatment was performed within 5 days before infusion, and CAR T cells were infused on day 0 (the dose was determined according to the requirements of climbing/expansion). The safety intensive observation period was 28 days after infusion, and the clinical efficacy after infusion was evaluated on days 28-34. The follow-up observation and evaluation were carried out according to the follow-up visit point, and the follow-up period was 1 year. From the second year, the telephone follow-up period was entered.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced solid tumors through histopathological diagnosis have a positive rate of ≥ 50% for mesothelin expression membrane and ≥ 50% for MUC1 expression in tumor tissue samples. PD-L1 expression is positive, and the sample source is within 2 years；
* Late stage malignant solid tumor patients who have failed standard treatment or are intolerant to such treatment and do not have a standard effective treatment plan ；
* Greater than or equal to 18 years of age and less than or equal to 70 years of age on day of signing informed consent；
* Life expectancy >3 months；
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；
* Satisfactory organ and bone marrow function as defined by the following：

  1. absolute neutrophil count must be greater than ≥ 1.5×10^9/L, lymphocyte count must be greater than ≥ 0.5×10^9/L, platelets must be greater than ≥ 90×10^9/L, hemoglobin must be greater than ≥ 90g/L without transfusion within 7 days or dependency on EPO;
  2. Total bilirubin must be less than or equal to two times (≤2.0x) the institutional normal upper limit; transaminases, serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST), must be less than or equal to 2.5 times (≤2.5x) the institutional normal upper limit (≤5x if there is hepatic metastasis);
  3. International normalized ratio (INR) or the PT is not greater than one and one half times (≤ 1.5) the upper limit of normal;
  4. Lung function: ≤ CTCAE grade 1 dyspnea and SaO2≥ 91%；
  5. Cardiac function: cardiac ejection fraction (LVEF) must be greater than fifty percent (≥50%) by echocardiogram or MUGA one month before enrollment.
* Subjects must have measureable disease as defined by RECIST 1.1 criteria;
* Subjects sufficiently understand the trial and willingly sign the informed consent；
* Male and Female subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for at least 12 months following the last dose of the study cell infusion and until no CAR-T cells can be detected after two consecutive PCR tests.

Exclusion Criteria:

* Subjects who have undergone other anti-tumor treatments (including radiation therapy, chemotherapy, small molecule, biological or immunotherapy, and other study drugs) other than lymphocytes depletion allowed by the protocol within one month prior to CAR-T infusion;
* Prior therapy with any gene therapy (including CAR-T cell therapy) or any T cell therapy home and abroad;
* Pregnant or breastfeeding women;
* Positive serological reactions for HIV and syphilis; Hepatitis B surface antigen positive, hepatitis B core antibody positive, and hepatitis B virus DNA copy number higher than the detection limit and/or greater than or equal to 1000 copies/mL; Or Hepatitis C virus infected individuals;
* Any uncontrollable active infection, coagulation disorders, or any other major illness;
* Patients with autoimmune diseases, organ transplantation and other immune related diseases under treatment, or long-term use of immunosuppressive drugs such as glucocorticoids: a. Glucocorticoids: users cannot stop using CAR-T cells 72 hours before infusion; b. Immunosuppressants other than glucocorticoids cannot be stopped ≥ 4 weeks before enrollment;
* History of severe cardiac or pulmonary disease, including hypertension that cannot be controlled by medication, and any of the conditions occurred within the past 6 months: congestive heart failure (New York Heart Association functional classification ≥3), cardiac angioplasty and stents, myocardial infarction, unstable angina, or other clinically significant heart disease;
* Detectable clinically relevant central nervous system (CNS) metastases and/or pathology such as epilepsy/seizure, brain Ischemia/ hemorrhage, dementia, cerebellar disease, or autoimmune disease affecting central nervous system.
* Patients at high risk of causing bleeding or perforation;
* Patients who had undergone major surgical procedures or significant trauma within 4 weeks before apheresis, or who were expected to require major surgery during the study period;
* Patient has a known history of a hematologic malignancy, or of another malignant primary solid tumor concurrently, with the exception of :Patients with in situ cervical cancer or breast cancer with no evidence of disease for ≥ 3 years after curative treatments;Patients who underwent successful definitive resection of in situ cancer with no evidence of disease for ≥5 years;
* Other circumstances that were deemed by the investigator to be inappropriate for trial participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2027-03-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | After 28 days of infusion
  Safety

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | After 28 days of infusion
  Tolerability
Objective response rate (ORR) | Month 12
  Clinical response will be assessed by RECIST 1.1
Progression-free survival (PFS) | Month 12
  PFS of patients receiving Fast CAR T cells
Overall survival (OS) | Month 12
  OS of patients receiving Fast CAR T cells
Peak Plasma Concentration (Cmax) | Month 12
  Pharmacokinetics (PK)
AUC | Day 28
  Pharmacokinetics (PK)
Pharmacodynamics (PD) | Day 28
  D of IL-2, IL-4, IL-6, IL-8, IL-10, IL-15, IFN-γ, TNF-α and MCP1 will be analysed after CAR T cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jinxing Lou, Principal Investigator — Shanghai Mengchao Cancer Hospital
Locations (1):
- Shanghai Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China